CLINICAL TRIAL: NCT04293471
Title: Prediction of Heart-failure and Mortality by Echocardiographic Parameters and Machine Learning in Individuals With Left Bundle Branch Block
Brief Title: Prediction of Outcome by Echocardiography in Left Bundle Branch Block
Acronym: EchoLBBB
Status: Recruiting | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Collaborators: Oslo University Hospital (Other); University of Bergen (Other); Norwegian University of Science and Technology (Other); University of Tromso (Other); KU Leuven (Other)
Responsible Party: Principal Investigator, Assami Rosner, MD PhD, University Hospital of North Norway
Other Study IDs: REK2019/134
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Left Bundle-Branch Block
Keywords: Left bundle branch block; strain-imaging; myocardial work assessment; machine learning
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with left bundle branch block have an increased risk for the development of heart-failure and death. However, risk factors for unfavorable outcomes are still poorly defined. This study aims to identify echocardiographic parameters and ECG characteristics by machine learning in order to develop individual risk assessment

DETAILED DESCRIPTION:
The project investigates patients with left bundle branch block (LBBB) which describes a specific block in the electrical conduction system, where the electrical impulses must follow a detour, with the result that different parts of the heart-muscle do not contract at the same time. This condition is called left ventricular dyssynchrony. LBBB can be found in people who are otherwise completely healthy and need not have any practical consequences. In others LBBB is present in patients with different heart diseases such as after myocardial infarctions or other diseases involving the heart-muscle. Patients with implanted pacemakers have a similar failure in the conduction system. Both conditions can increase the risk for development of heart-failure and cardiovascular death. Dyssynchrony can be treated with a special pacemaker (cardiac resynchronisation therapy, CRT) in addition to regular medical treatment. The therapy is well established and has shown to reduce morbidity and mortality and even reverse heart-failure in some patients completely. However, the patients in need and responding to CRT treatment is still not optimally defined. New echocardiographic parameters based on strain imaging such as regional myocardial work are able quantify the degree of dyssynchrony and give new insights into the interplay of activation delay through the LBBB and loading conditions and weakness of the myocardium due to other diseases. These new and complex measures can be integrated with clinical information by machine learning (ML) as a promising tools for accurate patient selection for CRT. The project aims to find markers on ultrasound improved by ML based selection to distinguish those patients who have problems associated with the branch block from those who remain stable. This will facilitate both, an optimized patient selection for CRT treatment and follow-up schedule for those who have a stable condition.

ELIGIBILITY:
Inclusion Criteria:

* QRS complex >130 ms and R-wave duration in
* V6 >70 ms
* ventricular pacing>50%
* Previously implanted cardiac resynchronisation therapy (CRT)

Exclusion Criteria:

* Typical right bundle branch block.
* No ability to give informed consent,
* non-cardiovascular co-mobidities with reduced life-expectancy < 1 year
* patients with complex congenital heart disease.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited based on epidemiological studies from Tromsø, where LBBB or ventricular pacing has been identified. Further in-hospital patients and patients from the out-patient clinics will be recruited due to ECG assessment
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death | 15 years
  Timepoint (day) of death and its cause
Death of any cause | 15 years
  Timepoint (day) of death and its cause

SECONDARY OUTCOMES:
Hospital admission due to heart-failure | 15 years
  Time point of hospital admission and main-diagnosis

OTHER OUTCOMES:
Remodelling | 5 years
  Increase or decrease of ventricular volume in ml
Cardiac function | 5 years
  Increase or decrease of ejection fraction in %
Heart failure | 5 years
  Increase or decrease of heart failure by proBNP and NYHA class

CONTACTS AND LOCATIONS:
Overall Officials: Assami Rösner, MD,PhD, Principal Investigator — University Hospital North Norway
Locations (1):
- University Hospital North Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: Yes
All individual analytic codes for participants fom other Norwegian Hospitals need to be transferred to University Hospital North Norway (UNN) for registering outcome follow-up
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: 15 years
Access Criteria: Patient have been included and five-year outcome data will have been revised.

DOCUMENTS (1):
  • Study Protocol (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT04293471/Prot_000.pdf